CLINICAL TRIAL: NCT06287580
Title: Antihypertensive Drug Effects on Cerebral Hemodynamics and Sympathetic Control in Older Hypertensive Patients
Brief Title: Effects of Antihypertensive Drug Treatment on Brain Blood Flow, Cognition, and Regulation of Nervous System in Older Adults With Hypertension.
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Takuro Washio, Post Doctoral Research Fellow- Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STU-2024-0140
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Essential Hypertension; Older Adults
Keywords: antihypertensive drug; cerebral blood flow; cognitive function
MeSH Terms: conditions — Essential Hypertension | interventions — Chlorthalidone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Antihypertensive drug treatment Arm (Active Comparator): Participants will take a fixed dose of chlorthalidone (a diuretic, 12.5 mg or 25 mg orally once daily) for one to two week, with study visits for laboratory assessment at before and after intervention.
  Interventions: Drug: chlorthalidone
- Placebo treatment Arm (Placebo Comparator): Participants will receive placebo treatment for one to two weeks, with study visits for laboratory assessment at before and after intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: chlorthalidone — chlorthalidone, 12.5 mg or 25 mg orally once daily
  Arms: Antihypertensive drug treatment Arm
Other: Placebo — Placebo tablet taken orally once daily
  Arms: Placebo treatment Arm

SUMMARY:
High blood pressure (BP) is a public health problem worldwide. Nearly three-quarters of older adults (age ~60 years) in the United States have high BP. High BP links to many health problems, like stroke. Drug treatments are typically used in clinics to reduce high BP and the risk of associated health problems. However, these drug treatments may not always benefit brain health. For example, drug treatment may reduce brain blood flow, which may reduce cognitive function in older adults with high BP. Alternatively, reduced brain blood flow may cause high BP due to increased nervous system activity (the so-called "fight or flight response"). Thus, monitoring brain blood flow may help to manage high BP during drug treatment.

It is unknown if brain blood flow and its control will be altered by drug treatment in older high BP patients. Therefore, study team will recruit older adults with high BP, who receive either drug treatment or a placebo for 1 to 2 weeks and will assess brain blood flow, cognitive function, and nervous system control before and after treatment.

Results from this study will provide novel and clinically relevant information on the impact of drug treatment for high BP on brain health. Investigators expect these results will suggest that it is crucial to measure brain blood flow, which may be a therapeutic new target for BP control and brain health.

ELIGIBILITY:
Inclusion Criteria:

* Older men and women with prehypertension or mild-to-moderate essential hypertension (clinic systolic blood pressure 120-169 and/or diastolic blood pressure 80-109 mmHg).

Exclusion Criteria:

* Any evidence of cardiovascular or pulmonary disease by medical history or by physical examination
* Severe hypertension (systolic BP ≥170 and/or diastolic BP ≥110 mmHg; for safety reasons) or secondary hypertension
* Being on ≥3 antihypertensive agents
* Chronic kidney disease (an estimated glomerular filtration rate >45 mL/min) or renal failure
* Diabetes mellitus (fasting glucose ≥126 mg/dL or 2-hour oral glucose tolerance test, glucose level ≥200 mg/dL) or other systemic illness
* Any history of substance abuse (other than tobacco)
* Current cigarette smokers
* History of gouty arthritis
* Taking hormonal replacement therapy
* Endurance-trained athletes
* Diagnosed Alzheimer's disease and related dementias

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in Muscle sympathetic nerve activity (MSNA) from baseline at post intervention | Baseline, post intervention
  Muscle sympathetic nerve activity will be measured using microneurography at the peroneal nerve. Muscle sympathetic nerve activity will be quantified by identification and measurement of sympathetic bursts in the integrated neurogram and expressed as burst frequency (mean number of bursts per unit time)
Change in cognitive performance from baseline at post intervention via Stroop Color and Word Test | Baseline, post intervention
  Change in cognitive performance is measured by Stroop Color and Word Test. Accuracy and reaction time in the Stroop Color and Word test are computed to assess cognitive performance.
Change in Cerebral blood flow from baseline at post intervention | Baseline, post intervention
  A probe will be placed over an artery in participant's neck and temple. Total cerebral blood flow is calculated as a sum of blood flow from the four arteries of the internal carotid artery and vertebral artery. The distribution of cardiac output to the brain is calculated as the percentage of total cerebral blood flow to cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: TAKURO WASHIO, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No